CLINICAL TRIAL: NCT06605196
Title: Improving Cancer Prevention and Control Through Academic-local Public Health Department Partnerships
Acronym: AHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R37CA262011 (NIH); R37CA262011 (NIH)
Record Dates: First submitted 2023-12-06; First posted 2024-09-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: Improving cancer prevention and control; academic-local public health department partnerships
MeSH Terms: conditions — Neoplasms | interventions — Health Resources

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation Arm (Experimental): The implementation arm will receive tailored, guided support to improve their AHD partnerships.
  Interventions: Behavioral: Resources and guided facilitation
- Control Arm (Active Comparator): The control arm will be referred to existing resources in the Learning Community but will not receive new resources or guided facilitation.
  Interventions: Behavioral: Existing resources

INTERVENTIONS:
Behavioral: Resources and guided facilitation — Participants in the intervention arm will participate in a planning period at the beginning of the intervention period to establish the goals for the partnership. The investigators will use the prioritized list of AHD partnership features developed in prior research to guide the initial planning period and then assist the partnership members to plan to implement the corresponding strategies focused on their areas of interest (e.g., developing collaborative projects, hiring faculty, staff, or students to conduct data analysis). The investigators will use telephone, email communication, and video conferencing to communicate with AHD partnerships, regularly assess progress towards goals, and adjust goals and strategies based on the progress. One additional in person visit to each AHD partnership in the intervention arm will be made in year 2 of implementation to review goals and progress and provide additional guidance and tailored support as needed.
  Arms: Implementation Arm
Behavioral: Existing resources — Individuals will be referred to existing resources in the Learning Community.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to understand how to leverage structures and processes of academic health department (AHD) partnerships to facilitate implementation of cancer related evidence-based programs and policies (EBPPs).

DETAILED DESCRIPTION:
The investigators will conduct a group-randomized study (total N=28 AHD partnerships) to evaluate the effect of strategies to increase implementation of cancer control and prevention EBPPs by supporting AHD partnerships. Partnerships will be randomized 1:1 to either an active implementation arm in which they will receive tailored strategies based on prior knowledge of successful partnerships or to an existing set of resources for AHD partnerships. A mixed methods approach will be used to evaluate changes in AHD partnerships and understand how contextual factors may have impacted the AHD partnership's ability to support EBPP adoption.

ELIGIBILITY:
Inclusion Criteria:

* Local health department practitioners who are involved in the implementation of cancer prevention and control programs within their communities and are engaged in an academic-health department partnership.
* Employees in academic settings currently partnering with local health departments. These partnerships could be located anywhere within the United States.

Exclusion Criteria:

• Individuals under the age of 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Evidence-Based Interventions | Baseline, 2 years post baseline
  Participants will see 5 questions about interventions related to specific public health program areas. They will be asked if their agency or institution has delivered those interventions within the last year. Possible score of 0 to 5. Higher score indicates a better outcome.
Academic Health Department Evidence-Based Interventions | Baseline, 2 years post baseline
  Participants will see 5 questions about interventions related to specific public health program areas. They will be asked if their academic health department has delivered those interventions within the last year. Possible score of 0 to 5. Higher score indicates a better outcome.

SECONDARY OUTCOMES:
Organizational Collaboration - Aligning strategy | Baseline, 2 years post baseline
  Survey participants will be asked to rate their perceptions of their academic-health department partnership on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Overall, the members of our academic local health department partnership...
  1. Work together to identify unmet needs in the community
  2. Work together to decide how to fill gaps in services and programs
  3. Act toward a common goal
  4. Are often in competition with one another (item reversed scored)
  5. Have trouble communicating (item reversed scored)
Organizational Collaboration - Coordinating Current Work | Baseline, 2 years post baseline
  Survey participants will be asked to rate their perceptions of their academic-health department partnership on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Overall, the members of our academic local health department partnership...
  1. Get a lot accomplished by working together
  2. Have trusting relationships
  3. Have access to resources that support collaboration between our organizations (e.g., expertise, facilities, funding)
  4. Keep each other up to date about the issues we work on
  5. Share information that helps public health practice work better
Joint Decision Making | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their academic-health department partnership on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with the following statements about your academic local health department partnership.
  1. Our partner organization(s) highly value the opinions of other organizations, including our own
  2. Within our partnership, we brainstorm together to find solutions to address problems facing the collaboration
  3. We work through differences to arrive at win-win solutions
Joint Operation | Baseline, 2 years post baseline
  Survey participants will be asked to rate their perceptions of their academic-health department partnership on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." An overall operation score will be calculated by taking the average of the 2 characteristics. Higher scores indicate stronger partnerships.
  Overall, the members of our academic local health department partnership...
  1. Have clearly defined roles and responsibilities
  2. Coordinate tasks well
Reduced Autonomy | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their academic-health department partnership on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Lower scores indicate a better outcome.
  Please indicate the extent to which you agree with the following statements about your academic local health department partnership.
  1. This partnership hinders our organization from meeting its own missions
  2. This partnership reduces our organization's independence
  3. This partnership brings about conflicting expectations
Resource Sharing | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their academic-health department partnership on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with the following statements about your academic local health department partnership.
  1. Within the partnership, we combine resources (e.g., financial, personnel, physical spaces)
  2. Within the partnership, we share information
  3. Within the partnership, we appreciate each other's contributions
Perceived Collaboration Outcomes | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their academic-health department partnership on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Our academic local health department partnership…
  1. increases mutual respect and trust between the organizations.
  2. fosters a shared understanding of the public health needs in our community and the effective ways to address these needs.
  3. increases the number of connections between individuals in each organization or with other organizations.
  4. fosters equal influence and power in decision-making among partners
  5. improves the health of our community.
  6. improves practice-informed teaching.
  7. improves research-informed practice.
  8. improves students' application of theory to practice.
Awareness of Evidence-Based Decision Making Culture Supportive of Evidence-Based Decision Making | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of opportunities to learn about and apply evidence-based decision making on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with the following statements.
  1. I am provided the time to identify evidence-based programs and practices.
  2. My direct supervisor recognizes the value of management practices that facilitate evidence-based decision-making
  3. My agency offers employees opportunities to attend evidence-based decision-making
Capacity and Expectations for Evidence-based Decision Making | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of opportunities to learn about and apply evidence-based decision making on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." Possible scores 1 to 5. Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with the following statements.
  1. Top leadership in my agency encourages use of evidence-based decision-making
Resource Availability | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of resource availability in their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with the following statements.
  1. Informational resources are available to my work group/division to promote the use of evidence-based decision-making
  2. My agency engages health organizations in a network of partners that share resources to facilitate evidence-based decision-making
  3. Stable funding is available for evidence-based decision-making
Evaluation Capacity | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of evaluation capacity in their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with the following statements.
  1. My agency plans for evaluation of interventions prior to implementation.
  2. My agency uses evaluation data to monitor and improve interventions.
  3. My agency distributes intervention evaluation findings to other organizations that can use our findings.
Individual Skills | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their individual public health skills on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." Scores for each of the 6 characteristics will be dichotomized into strongly agree/agree (1) and neither disagree or agree/disagree/strongly disagree (0). Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with each statement.
  1. I am knowledgeable about evidence-based public health processes.
  2. I have the skills I need to adapt evidence-based interventions from one population to another.
  3. I have the ability to lead efforts in evidence-based public health in my organization.
  4. I feel competent to manage change within my organization.
  5. I have the skills to effectively communicate information on evidence-based interventions to leaders in my organization.
  6. I have the skills to effectively communicate information on evidence-based interventions to decision make
Organizational Capacity for Evidence-Based Decision Making/Leadership | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of leadership in their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." Scores for each of the 7 characteristics will be dichotomized into strongly agree/agree (1) and neither disagree or agree/disagree/strongly disagree (0). Higher scores indicate a better outcome.
  1. Has developed a plan to facilitate implementation of evidence-based interventions.
  2. Has removed obstacles to the implementation of evidence-based interventions.
  3. Recognizes and appreciates employee efforts toward successful implementation of evidence-based interventions.
  4. Encourages planning for sustainability of programs.
  5. Perseveres through the ups and downs of implementing evidence-based interventions.
  6. Supports employees 'efforts to use evidence-based interventions.
  7. Reacts to critical issues regarding the implementation of evidence-based interventions by openly and effectively addressing the problem
Individual Skills for Health Equity | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of health equity within their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  Please indicate the extent to which you agree with each statement.
  1. I can describe how my work advances health equity.
  2. I can describe the causes of health inequities.
  3. I can describe health disparities among the populations in the communities I serve.
  4. I can identify ways to use evidence-based decision making to advance health equity.
  5. I can identify policies that will affect the social determinants of health and improve equity.
Leadership | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of leadership in their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." Scores for each of the 7 characteristics will be dichotomized into strongly agree/agree (1) and neither disagree or agree/disagree/strongly disagree (0).
  Leadership in my agency....
  1. Has developed a plan to facilitate implementation of evidence-based interventions.
  2. Has removed obstacles to the implementation of evidence-based interventions.
  3. Recognizes and appreciates employee efforts toward successful implementation of evidence-based interventions.
  4. Encourages planning for sustainability of programs.
  5. Perseveres through the ups and downs of implementing evidence-based interventions.
  6. Supports employees' efforts to use evidence-based interventions.
  7. Reacts to critical issues regarding the implementation of evidence-based interventions by openly and effectively addressing the problem.
Organizational Climate and Culture | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of organizational climate and culture within their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores mean a better outcome.
Organizational Characteristics Related to Health Equity | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of organizational climate and culture within their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." A summary score will be created as an average of the items within the domain. Possible scores 1 to 5. Higher scores indicate a better outcome.
  1. My agency adapts approaches to populations experiencing disparities
  2. My agency allows employees to dedicate time for addressing health equity (HE)
  3. Programs and policies in my agency are designed to improve HE
  4. My agency has systems in place to track our progress in addressing HE
  5. HE is a core value within my agency
  6. My agency is intentional about hiring staff members who represent communities experiencing inequities
  7. Leaders in my agency prioritize HE when implementing programs and policies
  8. Leaders in my agency place a high value on addressing HE
  9. HE is explicitly stated as a shared priority in collaborations w/ internal agency partners
Environmental Support | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." An overall environmental support score will be calculated by taking the average of the 3 characteristics. Possible score of 1 to 5. Higher score indicates a better outcome.
  For each statement, select the option that best indicates the extent to which you agree with the following statements about your agency.
  1. My agency has leadership support from outside of the agency (e.g., support from the governor or other elected officials)
  2. My agency and its work have strong public support (e.g., support from individuals in the community)
  3. My agency collaborates with sectors outside of health (e.g., business, parks and recreation programs, architecture).
Funding Stability | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." An overall funding stability score will be calculated by taking the average of the 5 characteristics. Possible score of 1 to 5. Higher score indicates a better outcome.
  For each statement, select the option that best indicates the extent to which you agree with the following statements about your agency.
  1. My agency's work exists in a supportive state economic climate.
  2. My agency implements policies to help ensure sustained funding.
  3. My agency is funded through a variety of sources.
  4. My agency has a combination of stable and flexible funding.
  5. My agency has sustained funding.
Strategic Planning | Baseline, 2 years post baseline
  Participants will be asked to rate their perceptions of their agency on a 5-point ordered scale from "Strongly disagree" to "Strongly agree." An overall strategic planning score will be calculated by taking the average of the 3 characteristics. Possible score of 1 to 5. Higher score indicates a better outcome.
  For each statement, select the option that best indicates the extent to which you agree with the following statements about your agency.
  1. My agency plans for future resource needs.
  2. My agency has a long-term financial plan.
  3. My agency has a sustainability plan.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Mazzucca-Ragan, Principal Investigator — Washington University School of Medicine
Locations (1):
- Prevention Research Center at Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Publications and underlying primary data generated as part of the proposed work will be shared. Publications will be made immediately available to the public without any embargo period.
Access Criteria: Electronic copies of publications will be deposited in PubMed Central using proper tagging of metadata to ensure online discoverability and accessibility within four weeks of acceptance by a journal. Underlying primary data (i.e., all survey- and qualitative data collected within grant activities) will be de-identified according to the Department of Health and Human Services (HHS) Regulations for the Protection of Human Subjects and Health Insurance Portability and Accountability Act (HIPAA) Privacy Rule and will be reviewed by our Institutional Review Board. De-identified data will be standardized and placed in a data repository that the investigators will develop for data sharing with a broader research community in a timely manner. The data repository will be updated upon publication of manuscripts. No limitations to the immediate and broad release of publication and underlying primary data are anticipated,

REFERENCES:
- [Derived] Mazzucca-Ragan S, Allen P, Amos K, Barker AR, Brewer M, Erwin PC, Gannon J, Gao F, Jacob RR, Lengnick-Hall R, Brownson RC. Improving cancer prevention and control through implementing academic-local public health department partnerships - protocol for a cluster-randomized implementation trial using a positive deviance approach. Implement Sci Commun. 2025 Feb 24;6(1):20. doi: 10.1186/s43058-025-00706-z. PMID 39994666
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu